CLINICAL TRIAL: NCT00400413
Title: Phonological Perception and Learning to Read : the Neuroanatomy of Reading in Congenitally Deaf Persons
Brief Title: Neuroanatomy of Reading in Congenital Deafness.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other); Conseil Régional d'Alsace (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2865
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Congenital Deafness
Keywords: Neuropsychology; fMRI; Reading; Phonology; Deafness
MeSH Terms: conditions — Deafness

INTERVENTIONS:
Procedure: fMRI

SUMMARY:
The aim of the research is to investigate phonological processing in deafness and to examine its influence on the neuroanatomy of reading.The basic hypothesis is that insofar as the ability to read is closely related to the ability to segment and represent speech units, the neuroanatomy of reading in deaf would be different from the one of hearing readers.

ELIGIBILITY:
Inclusion criteria:

* adult
* full education

Exclusion criteria:

* reading impairment
* fMRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-11 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noëlle Metz-Lutz, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Clinique Neurologique - Hôpital Civil, Strasbourg, France

REFERENCES:
- [Result] Aparicio M, Gounot D, Demont E, Metz-Lutz MN. Phonological processing in relation to reading: an fMRI study in deaf readers. Neuroimage. 2007 Apr 15;35(3):1303-16. doi: 10.1016/j.neuroimage.2006.12.046. Epub 2007 Jan 25. PMID 17329129